CLINICAL TRIAL: NCT00267137
Title: Study for Atrial Fibrillation Reduction (SAFARI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation, Bradycardia
Keywords: Pacemaker, Atrial Fibrillation/Therapy
MeSH Terms: conditions — Atrial Fibrillation; Bradycardia

INTERVENTIONS:
Device: Pacing Algorithms

SUMMARY:
Atrial fibrillation (AF), which is the name for rapid beats in the upper chambers of the heart, is the world's most common kind of irregular heart beat. People with AF experience symptoms such as heart palpitations (a racing or pounding feeling in the chest), shortness of breath, dizziness, fatigue or weakness. Although AF can occur in otherwise healthy people for no apparent reason, it is sometimes associated with high blood pressure, heart disease or lung problems. The purpose of the SAFARI trial is to study the effectiveness of pacing algorithms in the upper chamber of the heart for patients who have both AF and bradycardia (slow heart beat).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a slow heartbeat who are in need of dual chamber pacing (pacing in both the atrium and ventricle).
* Subjects who have experienced at least two episodes of rapid heart beats three months prior to enrollment.

Exclusion Criteria:

* Subjects who have a history of permanent (chronic) or persistent (non self-terminating) atrial fibrillation.
* Subjects with atrial fibrillation due to reversible cause, (e.g. thyroid disease, pericarditis, post-surgery, alcohol abuse).
* Subjects with a history of one or more cardioversions (changing an abnormal heart rhythm into a normal one by either using medication or by the application of an electric shock) six months prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 540
Dates: Start 2002-09 (Actual); Primary Completion 2005-09-11 (Actual); Study Completion 2006-07-21 (Actual)

PRIMARY OUTCOMES:
Safety/Efficacy

SECONDARY OUTCOMES:
Various

CONTACTS AND LOCATIONS:
Overall Officials: Not Required For IDE Studies
Locations (34):
- United States (34):
  - Yuma, Arizona
  - Fayetteville, Arkansas
  - Fort Smith, Arkansas
  - Bakersfield, California
  - Berkeley, California
  - Los Angeles, California
  - Aurora, Colorado
  - Stamford, Connecticut
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Ormond Beach, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lombard, Illinois
  - Springfield, Illinois
  - Shreveport, Louisiana
  - Brighton, Massachusetts
  - Lansing, Michigan
  - Saint Paul, Minnesota
  - Paterson, New Jersey
  - Ridgewood, New Jersey
  - East Syracuse, New York
  - Rochester, New York
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Elyria, Ohio
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Background] Gold MR, Hoffmann E; SAFARI Investigators. Rationale and design of a randomized clinical trial to assess the role of overdrive and triggered prevention pacing therapies in reducing atrial fibrillation: the Study of Atrial Fibrillation Reduction (SAFARI). Am Heart J. 2006 Aug;152(2):231-6. doi: 10.1016/j.ahj.2005.11.012. PMID 16875902